CLINICAL TRIAL: NCT03880344
Title: Randomized Control Trial Investigating the Effectiveness of Vibration Therapy on Sarcopenia in Osteoarthritis Knee Patients
Brief Title: Investigating the Effectiveness of Vibration Therapy on Sarcopenia in Osteoarthritis Knee Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Ho Ki Wai, Clinical Professional Consultant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CUHK_2018.403
Record Dates: First submitted 2019-03-06; First posted 2019-03-19 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Knee Arthropathy; Osteoarthritis, Knee; Knee Osteoarthritis
Keywords: vibration therapy; Knee Osteoarthritis; Knee Arthropathy
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibration Therapy + Normal Out-Patient Physiotherapy (Experimental): Patients' randomized to this group will receive vibration therapy as a pre-operative rehabilitation programme 3 times a week for 3 months. Regular out-patient department physiotherapy will also be given. They will be assessed 6 weeks and 6 months post operatively.
  Interventions: Device: Vibration Therapy; Combination Product: Physiotherapy
- Normal Out-Patient Department Physiotherapy (Active Comparator): Patients randomized to this group will receive regular out-patient department physiotherapy postoperatively for 6 months. They will be assessed 6 weeks and 6 months post operatively.
  Interventions: Combination Product: Physiotherapy

INTERVENTIONS:
Device: Vibration Therapy — Vibration therapy as a pre-operative rehabilitation programme 3 times a week for 3 months + Normal Regular out-patient department physiotherapy
  Arms: Vibration Therapy + Normal Out-Patient Physiotherapy
Combination Product: Physiotherapy — Physiotherapy as post-operative rehabilitation programme for 6 months.

SUMMARY:
Osteoarthritis (OA) is one of the commonest chronic degenerative conditions affecting our aging population. It limits joint movement and causing disability in elderlies due to discordant symptoms such as pain and stiffness. The prevalence of radiologic knee osteoarthritis increases in proportion to age, reaching an astounding 64.1% for patients whom are over 60 years of age. In addition the prevalence of symptomatic knee OA has been shown to be around 10% in people who are 60 years and older.

DETAILED DESCRIPTION:
Patients with end stage OA often adopt a sedentary lifestyle causing mobility and functionality decline to avoid joint pain and stiffness. This dysfunctions a series of antioxidant response cascades which eventually leads to muscle atrophy of the knee. Notably, muscle atrophy and weakness (i.e. sarcopenia) often accompanies with OA. However the relationship between these symptoms and OA remains undefined and no strong consensus have been made thus far. Our ongoing longitudinal study on muscle strength and functionality which investigates the prevalence of sarcopenia in end stage OA patient's pre and post operation (Total Knee Replacement) have reflected that 24% with severe knee OA patients also suffered sarcopenia. In addition, these patients also showed a much slower recovery and longer length of stay in hospital after undergoing surgical operation.

The effect of clinical sarcopenia affects our locomotion system in the aging population. Weakness in patients and decline in muscle strength results in significant functional impairment are often seen in the cohort, leading to fragility, falls, fractures and disability.

Many authors have tried to explain the pathophysiology of sarcopenia in an attempt to link the disorder to a molecular or biochemical level in numerous literature. Satellite cells (a myogenic stem cell), Insulin like growth factor 1 (IGF-1) (an important mediator of muscle growth and regeneration affecting muscle function) and fast twitch muscle fibres are three major molecular composites that have been widely studied. Evidence have suggested the close relationship between them and muscle atrophy and weakness. However, these studies have either shown the results from an animal standpoint or they lack specificity and further research is necessary to confirm their role in patients suffering from sarcopenia.

Attempts have also been made to discover the most effective intervention to treat or even eliminate the chances of sarcopenia. Among these studies resistance exercises have been documented the most.

Evidence showed that progressive resistance and aerobic exercises are most beneficial for the prevention and treatment of sarcopenia. Resistant training that such as lifting weights, strength resistance bands, resistance machines has shown to improve protein synthesis in skeletal muscle cells leading to better muscle strength and mass, leading to muscle hypertrophy and promotes muscle power. Our previous knowledge transfer study on developing an aerobic exercise (i.e. Tai Chi Exercise) for end stage OA patients also showed similar positive effects in subjects, decreasing their pain and stiffness symptoms and limitations in physical activity. Though resistance exercise showed promising effects, are safe and strongly advised interventions based on documented and our previous study, the elderly populations often accompanies with other physical symptoms (such as back pain) and diminished fine motor skills that may limit their range of movement in these exercise regimes. In addition, resistive exercises are extremely technical and is essential to execute with proper form to avoid further injury; hence these exercises are unable to perform safely alone at home, making the intervention less autonomous.

Vibration therapy is a noninvasive biophysical modality and has been demonstrated in a number of studies showing multiple positive effects in terms of postural control, balancing ability, circulation and most importantly muscle strength. Two of our previous studies investigated the long term effects on muscle performance and bone quality in using low-magnitude high frequency vibration. Though the results showed that the treatment is an effective method in fall prevention by improving on both frontiers, these two studies' main subject focuses were on the elderly population as a whole. A study pivoting on subjects with co-existing diagnosis of sarcopenia and OA is crucial to investigate the effectiveness of this therapy method. Limited studies have shown positive effects of vibration therapy on osteoarthritis, however, these studies were limited to a single gender (i.e. females) or contained subject recruitment bias or assessment period of less than 6 months. A randomized control trial with a longer assessment period is essential to investigate the true effects of vibration therapy on knee OA patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged over 45 with end stage knee OA
* Patient has been scheduled for TKR
* Able to comply with the assessments and has given oral and written consent

Exclusion Criteria:

* Patients with connective tissue disorders or myositis condition
* Previous cases of alcoholism or drug abuse
* Pregnancy or breast feeding

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee Flexion/Extension Strength | Baseline Assessment
  Muscle strength on the quadriceps is measured by instructing the patient to perform an active knee flexion/extension movement in a sitting position with both feet free from ground, and the hip and knee joint flexed at 90%. The optimal isometric force of the knee flexion/extension movement are measured by the dynamometer attached at the malleoli level with a strap. The measurements (0 to 30 cm) will be taken at maximum force for three times.
Knee Flexion/Extension Strength | Pre-Operative Assessment
  Muscle strength on the quadriceps is measured by instructing the patient to perform an active knee flexion/extension movement in a sitting position with both feet free from ground, and the hip and knee joint flexed at 90%. The optimal isometric force of the knee flexion/extension movement are measured by the dynamometer attached at the malleoli level with a strap. The measurements (0 to 30 cm) will be taken at maximum force for three times.
Knee Flexion/Extension Strength | Post-Operative 6 weeks
  Muscle strength on the quadriceps is measured by instructing the patient to perform an active knee flexion/extension movement in a sitting position with both feet free from ground, and the hip and knee joint flexed at 90%. The optimal isometric force of the knee flexion/extension movement are measured by the dynamometer attached at the malleoli level with a strap. The measurements (0 to 30 cm) will be taken at maximum force for three times.
Knee Flexion/Extension Strength | Post-Operative 6 months
  Muscle strength on the quadriceps is measured by instructing the patient to perform an active knee flexion/extension movement in a sitting position with both feet free from ground, and the hip and knee joint flexed at 90%. The optimal isometric force of the knee flexion/extension movement are measured by the dynamometer attached at the malleoli level with a strap. The measurements (0 to 30 cm) will be taken at maximum force for three times.
Knee Flexion/Extension Strength | Post-Operative 12 months
  Muscle strength on the quadriceps is measured by instructing the patient to perform an active knee flexion/extension movement in a sitting position with both feet free from ground, and the hip and knee joint flexed at 90%. The optimal isometric force of the knee flexion/extension movement are measured by the dynamometer attached at the malleoli level with a strap. The measurements (0 to 30 cm) will be taken at maximum force for three times.

SECONDARY OUTCOMES:
Whole body lean muscle mass | Baseline Assessment
  DXA measurement scan
Whole body lean muscle mass | Pre-Operative Assessment
  DXA measurement scan
Whole body lean muscle mass | Post-Operative 6 months
  DXA measurement scan
Muscle Biopsy | Intra-Operatively
  Types of muscle fibers and satellite cells as Assessed by Muscle Biopsy Assessment
Knee Functions measure by the Knee Society Score | Baseline Assessment
  Physician will assess on the Visual Analog Scale in pain score (None to Severe), Flexion Contracture (None to >20°), Extension lag (None to 20°), Total Range of Flexion (0-5° to 121-125°), Alignment (0° to Over 15°), Antero-posterior stability (<5mm to 10+mm), Mediolateral stability (<5° to 15°). Patients will record individuals' satisfaction, functional activities, and expectations.
Knee Functions measure by the Knee Society Score | Pre-Operative Assessment
  Physician will assess on the Visual Analog Scale in pain score (None to Severe), Flexion Contracture (None to >20°), Extension lag (None to 20°), Total Range of Flexion (0-5° to 121-125°), Alignment (0° to Over 15°), Antero-posterior stability (<5mm to 10+mm), Mediolateral stability (<5° to 15°). Patients will record individuals' satisfaction, functional activities, and expectations.
Knee Functions measure by the Knee Society Score | Post-Operative 6 weeks
  Physician will assess on the Visual Analog Scale in pain score (None to Severe), Flexion Contracture (None to >20°), Extension lag (None to 20°), Total Range of Flexion (0-5° to 121-125°), Alignment (0° to Over 15°), Antero-posterior stability (<5mm to 10+mm), Mediolateral stability (<5° to 15°). Patients will record individuals' satisfaction, functional activities, and expectations.
Knee Functions measure by the Knee Society Score | Post-Operative 6 months
  Physician will assess on the Visual Analog Scale in pain score (None to Severe), Flexion Contracture (None to >20°), Extension lag (None to 20°), Total Range of Flexion (0-5° to 121-125°), Alignment (0° to Over 15°), Antero-posterior stability (<5mm to 10+mm), Mediolateral stability (<5° to 15°). Patients will record individuals' satisfaction, functional activities, and expectations.
Knee Functions measure by the Knee Society Score | Post-Operative 12 months
  Physician will assess on the Visual Analog Scale in pain score (None to Severe), Flexion Contracture (None to >20°), Extension lag (None to 20°), Total Range of Flexion (0-5° to 121-125°), Alignment (0° to Over 15°), Antero-posterior stability (<5mm to 10+mm), Mediolateral stability (<5° to 15°). Patients will record individuals' satisfaction, functional activities, and expectations.
Knee Function measures by 6 meter Timed Walking Gait Test | Baseline Assessment
  The 10 meter timed walking test is a well-established and documented test for assessment for gait speed in patients. However, due to space limitations and the exhaustive nature of the test for patients with OA, the 6 meter test has been documented to be a valid and reliable substitute. Patients will be asked to walk a straight line of 6 meters where the time taken to complete the distance will be measured. (<7.5 seconds is normal).
Knee Function measures by 6 meter Timed Walking Gait Test | Pre-Operative Assessment
  The 10 meter timed walking test is a well-established and documented test for assessment for gait speed in patients. However, due to space limitations and the exhaustive nature of the test for patients with OA, the 6 meter test has been documented to be a valid and reliable substitute. Patients will be asked to walk a straight line of 6 meters where the time taken to complete the distance will be measured. (<7.5 seconds is normal).
Knee Function measures by 6 meter Timed Walking Gait Test | Post-Operative 6 weeks
  The 10 meter timed walking test is a well-established and documented test for assessment for gait speed in patients. However, due to space limitations and the exhaustive nature of the test for patients with OA, the 6 meter test has been documented to be a valid and reliable substitute. Patients will be asked to walk a straight line of 6 meters where the time taken to complete the distance will be measured. (<7.5 seconds is normal).
Knee Function measures by 6 meter Timed Walking Gait Test | Post-Operative 6 months
  The 10 meter timed walking test is a well-established and documented test for assessment for gait speed in patients. However, due to space limitations and the exhaustive nature of the test for patients with OA, the 6 meter test has been documented to be a valid and reliable substitute. Patients will be asked to walk a straight line of 6 meters where the time taken to complete the distance will be measured. (<7.5 seconds is normal).
SF-12 | Baseline Assessment
  The 36-Item Short Form Health Survey (SF-12) will be used to measure the health related Quality of Life. The SF-12 has twelve questions ; the scores are weighted sums of the questions in each section. Scores range from 0 - 60. Lower scores = more disability, higher scores = less disability.
SF-12 | Pre-Operative Assessment
  The 36-Item Short Form Health Survey (SF-12) will be used to measure the health related Quality of Life. The SF-12 has twelve questions ; the scores are weighted sums of the questions in each section. Scores range from 0 - 60. Lower scores = more disability, higher scores = less disability.
SF-12 | Post-Operative 6 weeks
  The 36-Item Short Form Health Survey (SF-12) will be used to measure the health related Quality of Life. The SF-12 has twelve questions ; the scores are weighted sums of the questions in each section. Scores range from 0 - 60. Lower scores = more disability, higher scores = less disability.
SF-12 | Post-Operative 6 months
  The 36-Item Short Form Health Survey (SF-12) will be used to measure the health related Quality of Life. The SF-12 has twelve questions ; the scores are weighted sums of the questions in each section. Scores range from 0 - 60. Lower scores = more disability, higher scores = less disability.
Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | Baseline Assessment
  The WOMAC will be used as a self-administered health status measure in assessing pain, stiffness, and function in patients with OA of the hip or knee. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | Pre-Operative Assessment
  The WOMAC will be used as a self-administered health status measure in assessing pain, stiffness, and function in patients with OA of the hip or knee. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | Post-Operative 6 weeks
  The WOMAC will be used as a self-administered health status measure in assessing pain, stiffness, and function in patients with OA of the hip or knee. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations. With a scale ranges from 0 to 96. Lower scores = more disability, higher scores = less disability.
Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | Post-Operative 6 months
  The WOMAC will be used as a self-administered health status measure in assessing pain, stiffness, and function in patients with OA of the hip or knee. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations. With a scale ranges from 0 to 96. Lower scores = more disability, higher scores = less disability.
IPAQ | Baseline Assessment
  The 36-Item Short Form Health Survey (SF-12) will be used to measure health-related physical activity (PA) performance. With a scale ranges from 0 to 96. Lower scores = more disability, higher scores = less disability.
IPAQ | Pre-Operative Assessment
  The 36-Item Short Form Health Survey (SF-12) will be used to measure health-related physical activity (PA) performance. Score is expressed as MET-min per week: MET level x minutes of activity x events per week. Computed to fall into the category of: "Low", "Moderate" and "High" level of Physical Activity.
IPAQ | Post-Operative 6 weeks
  The 36-Item Short Form Health Survey (SF-12) will be used to measure health-related physical activity (PA) performance. Score is expressed as MET-min per week: MET level x minutes of activity x events per week. Computed to fall into the category of: "Low", "Moderate" and "High" level of Physical Activity.
IPAQ | Post-Operative 6 months
  The 36-Item Short Form Health Survey (SF-12) will be used to measure health-related physical activity (PA) performance. Score is expressed as MET-min per week: MET level x minutes of activity x events per week. Computed to fall into the category of: "Low", "Moderate" and "High" level of Physical Activity.
Hand-grip Strength | Baseline Assessment
  Average of 3 times hand-grip strength values measures by a hand dynamometer grip strength meter.
Hand-grip Strength | Pre-Operative Assessment
  Average of 3 times hand-grip strength values measures by a hand dynamometer grip strength meter.
Hand-grip Strength | Post-Operative 6 weeks
  Average of 3 times hand-grip strength values measures by a hand dynamometer grip strength meter.
Hand-grip Strength | Post-Operative 6 months
  Average of 3 times hand-grip strength values measures by a hand dynamometer grip strength meter.
Gait Speed | Baseline Assessment
  6 meter timed walking gait test
Gait Speed | Pre-Operative Assessment
  6 meter timed walking gait test
Gait Speed | Post-Operative 6 weeks
  6 meter timed walking gait test
Gait Speed | Post-Operative 6 months
  6 meter timed walking gait test

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopaedics & Traumatology, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided